CLINICAL TRIAL: NCT03929991
Title: Maternal Cesarian Section Infection (MACSI) in Sierra Leone: an Observational Study
Brief Title: Maternal Cesarian Section Infection (MACSI) in Sierra Leone
Acronym: MACSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Doctors with Africa - CUAMM (Other)
Collaborators: University of Bari (Other); University of Palermo (Other)
Responsible Party: Sponsor
Other Study IDs: 1902
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Infection; Cesarean Section Complications; Site Infection; Maternal Death
Keywords: Site infection; Sierra Leone; Africa; Cesarean Infection; Maternal Mortality
MeSH Terms: conditions — Infections; Maternal Death | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: All women admitted or already hospitalized with suspected or confirmed infection after C/S will be screened for inclusion in the study as a case. Case confirmation will be clinically established by an infectious disease expert.SSI post C/S will be classified as:
  * Superficial incisional surgical site infection,
  * Deep incisional surgical site infection,
  * Organ/space surgical site infection.
  Interventions: Other: Observational
- Control: For each case, 3 patients undergoing the C/S on the same day and admitted to the same ward but not presenting Surgical Site Infection
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — To record social and clinical characteristics

SUMMARY:
Up to 1 in 5 women in Africa who deliver their baby by cesarean section get a wound infection.

Surgical site infections (SSIs) are largely preventable, but they represent a considerable burden for health-care systems, particularly in low-income and middle-income countries. The prevention of these infections is complex and requires the integration of a range of preventive measures before, during, and after surgery.

The aim of the proposed project is to determine the risk factors of Surgical Site Infection post-Cesarean Section in women admitted to Princess Christian Maternity Hospital (PCMH) in Freetown, Sierra Leone. Secondary aims are to determine the incidence of SSI and the predictors of a negative outcome in women with post-CS SSI.

DETAILED DESCRIPTION:
Rationale: More than 1 in 10 people who have surgery in low and middle-income countries (LMICs) get surgical site infection. People's risk of SSI in LMICs is 3 to 5 times higher than in high-income countries. Up to 1 in 5 women in Africa who deliver their baby by cesarean section get a wound infection.

Surgical site infections (SSIs) are largely preventable, but they represent a considerable burden for health-care systems, particularly in low-income and middle-income countries. The prevention of these infections is complex and requires the integration of a range of preventive measures before, during, and after surgery.

Objective: The aim of the proposed project is to determine the risk factors of Surgical Site Infection post-Cesarean Section in women admitted to Princess Christian Maternity Hospital (PCMH) in Freetown, Sierra Leone. Secondary aims are to determine the incidence of SSI and the predictors of a negative outcome in women with post-CS SSI.

Study design: This is a prospective case-control (1:3 ratio) study. Study population and Methods: All women admitted or already hospitalized with suspected or confirmed infection after C/S will be screened for inclusion in the study as a case. Case confirmation will be clinically established by an infectious disease expert. For each case, 3 patients undergoing the C/S on the same day and admitted to the same ward but not presenting SSI, will be selected as controls.

Sample size: No formal sample size calculation is performed.

Main study parameters/primary endpoints: SSI post C/S will be classified as:

Superficial incisional surgical site infection, Deep incisional surgical site infection; Organ/space surgical site infection Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Because all proceedings in the method of this study are based on common clinical practice, there are no serious adverse events (SAEs) expected.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women undergoing a C/S in on the hospitals during the study period will be eligible to participate in this study.

Exclusion Criteria:

The following conditions will not be considered as outcome, unless they present with systemic repercussion due to infection. For example:

* Vaginosis, candidiasis
* Lower tract urinary infection
* Fungal infections of the skin (athlete's foot, jockitch, ringworm, and yeast infections)
* Otitis
* Pharyngitis
* Herpes simplex, Herpes Zoster (Shingles)
* Uncomplicated chronic infection
* Sexually transmitted infections (Gonorrhoea, Syphilis, Trichomonas, Chlamydia, Hepatitis, HIV)
* Tuberculosis
* Bacterial colonization (presence of microorganisms without clinical signs/symptoms)
* Known vaginal, urethral and/or rectal GBS colonization
* Asymptomatic bacteriuria
* Known oropharyngeal colonization
* Non-infectious hypothermia/hyperthermia (e.g. related to epidural, thyroid storm, prostaglandin administration) during hospital stay

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All women admitted to Princess Christian Maternity Hospital (PCMH) in Freetown, Sierra Leone.
Study Population: Pregnant women undergoing a C/S in an urban tertiary referral maternity hospital PCMH, Freetown (population served: 1'500'000; n. of total deliveries in 2017: 6'861; number of C/S in 2017: 2'028 ).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence | From hospital admission to hospital discharge, an overage of 1 month
  To determine the incidence of SSI after CS at PCMH during the study period

SECONDARY OUTCOMES:
Prevalence of Main Features | From hospital admission to hospital discharge, an overage of 1 month
  To describe the main features of SSI after CS in women admitted at PCMH
Prevalence of Negative Outcome | From hospital admission to hospital discharge, an overage of 1 month
  To assess predictor of negative outcomes of SSI after CS
Screening of Risk factors | From hospital admission to hospital discharge, an overage of 1 month
  To determine the risk factors of Surgical Site Infection post Cesarean Section

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Putoto, PhD, Principal Investigator — Department of operational research Doctors with Africa CUAMM Padova, Italy
Locations (1):
- Princess Christian Maternity Hospital, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: Undecided